CLINICAL TRIAL: NCT06810102
Title: The Effect of the Bırth Process Watched to Nursıng Students Through Vırtual Realıty Glasses on the Students' Perceptıon of Traumatıc Bırth and Bırth Preferences
Brief Title: Vırtual Realıty Glasses' Traumatıc Bırth Perceptıon and Bırth Preferences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, NURDİLAN SENER, phd of woman health nursing, asoc prof., Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: fıratuniversty
Record Dates: First submitted 2024-12-20; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: NURSING STUDENTS
Keywords: birth preferences.; virtual reality glasses; perception of traumatic birth

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a randomized controlled experimental model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): Before the lesson, students will watch a video of the actual birth. The video is available on YouTube (https://www.youtube.com/watch?v=IRjOO6V83Uw) and was edited and voiced by the researcher to its final form. The video includes observations starting before birth, the birth itself and the early postpartum period.
  Interventions: Other: VIRTUAL REALITY GLASSES
- control (No Intervention): No intervention will be made

INTERVENTIONS:
Other: VIRTUAL REALITY GLASSES — There will be a video screening
  Arms: experimental

SUMMARY:
Birth is an irreplaceable experience in an individual's life, and can have critical health consequences for both the mother and the baby. Healthcare professionals, especially nurses, play an important role in the management, support and education of this process. Nursing students' knowledge and experience about labor is an important factor that affects both their professional development and future patient care.

Traditional education methods may have limited impact on healthcare professionals in learning about the birth process. Instead, the use of virtual reality (VR) technology offers students the opportunity to experience the birth process realistically. In a virtual reality environment, nursing students can understand the physiological stages of birth, its effects on the mother and baby, and the emotional aspects of the birth process more deeply. This has the potential to change traumatic perceptions of the birth process, and can also have an impact on birth preferences.

The perception of traumatic birth is shaped by individuals' negative thoughts and feelings about their birth experiences. These perceptions emerge as an important factor affecting future birth preferences and health care application status beyond the birth process. During nursing education, shaping these perceptions of students and providing them with positive experiences is of critical importance. Experiencing labor with virtual reality can reduce students' negative perceptions of birth and help them make more conscious choices about birth options.

DETAILED DESCRIPTION:
Birth is a natural and enjoyable process that includes surprises that do not go well. While nurses usually witness positive and uplifting births, they also encounter traumatic and upsetting events. Especially when faced with difficult births, this situation can have an intense psychological impact and a perception of traumatic birth can occur. Student nurses who provide care in delivery rooms during their training feel empathic feelings towards their fellow women when they encounter a traumatic event during birth and as a result, they become vulnerable to secondary traumatic stress. This situation can put students under a heavy psychological burden and increase their perception of traumatic birth . The perception of birth is the most important factor that causes a woman to have a wonderful experience or a negative birth story that she will remember for the rest of her life. Women's negative perception of birth causes an increase in the rates of interventional birth (oxytocin use, episiotomy and amniotomy practices) and elective cesarean section, and negatively affects birth preference and type, postpartum satisfaction, postpartum emotional process, family relationship and mother-baby bonding. The education process of nursing students is an important opportunity to change their existing negative perceptions of birth, increase their awareness of the issue and implement initiatives aimed at these. It is thought that nurses with a positive perception of birth will make more effective interventions in terms of reducing and encouraging the fears of the pregnant woman at every stage of birth. The ultimate goal of nursing education is to encourage the application of theoretical knowledge in clinical practice. However, limited clinical practice time affects students' opportunity to gain clinical experience with real patients. Due to the rapid development of information technology and the inadequacy of the nursing workforce, a transformation is needed in nursing education to prepare nursing students for evolving and complex healthcare environments. Virtual reality (VR) is a computer-generated three-dimensional graphical representation of a natural or imaginary environment into which users are immersed through a special headset or a series of screen walls. In general, VR can be a promising technology for enhancing learning through experiential learning . Educators in the field of women's health nursing face various challenges when trying to provide the best learning experience for students. Students are only in the role of observers rather than an active nursing role during the labor and delivery process. Accordingly, it is thought that the births they observe may affect their thoughts about birth . In this context, our study aimed to determine the effect of the labor process that nursing students watched through virtual reality glasses on the students' perception of traumatic birth and birth preferences.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Having taken a gynecology course

Exclusion Criteria:

* Having witnessed any labor before,
* Having any psychiatric diagnosis,
* Having any neurological disease (such as epilepsy) that will cause seizures,
* Having any diagnosis that causes dizziness in the patient, such as vertigo.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women's perception and preferences of childbirth
Enrollment: 109 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
traumatic perception of birth | 1 month
  It is thought that showing the birth process to nursing students through virtual reality will reduce the score they will receive on the traumatic birth perception scale and reduce the perception of traumatic birth.
Birth preferences | 1 month
  It is thought that by showing the birth process to nursing students in virtual reality, birth preferences will change and the rate of cesarean births will decrease.

CONTACTS AND LOCATIONS:
Locations (1):
- NURDİLAN, Elâzığ, Elâzığ, Turkey (Türkiye)